CLINICAL TRIAL: NCT00711282
Title: A Prospective, Randomized, Controlled Study to Evaluate Buccal Bone Preservation Using Fixture MicroThread™ OsseoSpeed™ Placed in Fresh Extraction Sockets the Maxilla.
Brief Title: Study of Bone Preservation When OsseoSpeed™ Implants Are Placed Immediately Following Tooth Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YA-OSS-0009
Record Dates: First submitted 2008-07-07; First posted 2008-07-08 (Estimated); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Jaw, Edentulous, Partially
Keywords: Replacement of non-restorable single tooth/teeth
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Device: OsseoSpeed™
- B (Experimental)
  Interventions: Device: OsseoSpeed™

INTERVENTIONS:
Device: OsseoSpeed™ — OsseoSpeed™ MicroThread™, diameters of 3.5 and 4.0 mm.
  Arms: A
Device: OsseoSpeed™ — OsseoSpeed™ MicroThread™, diameters of 4.5 and 5.0 mm.
  Arms: B

SUMMARY:
The purpose of this study is to evaluate the clinical performance of implants placed in individuals who are about to loose one or more of their upper teeth. The main objective is to study how the surrounding bone tissue reacts to two different shapes of implants. Clinical performance, in wider terms, means esthetics and long lasting function. Half of the patients will receive a cylindrically shaped implant and the other half will receive a conical-cylindrical implant. The implants will be placed and after a healing period of 16 weeks the gum will be re-opened and the bone tissue response clinically evaluated. Permanent artificial tooth/teeth will be attached six weeks after that.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* At least 18 years at inclusion
* At least 20 teeth with expected functional balanced occlusion after restoration
* In need of one or more implants replacing teeth to be removed in the maxilla within region 15 to 25
* Presence of an intact extraction socket following removal of the natural tooth defined by: (1) a situation where the marginal border of the facial bone crest deviates less than or equal to 2 mm from that of the expected normal anatomy of the site/region, (2) a marginal border of a potential facial fenestration at least 3 mm apical of the marginal bone crest
* Presence of an extraction socket anatomy, following removal of the natural tooth, suitable for both cylindrical and conical/cylindrical implants

Exclusion Criteria:

* Untreated rampant caries and uncontrolled periodontal disease
* Absence of adjacent (mesial and/or distal) natural tooth root
* Uncontrolled diabetes (subjects history does not reveal the absence of control of insulin-dependent / non-insulin dependent Diabetes Mellitus)
* Current alcohol or drug abuse
* Systemic or local disease or condition that would compromise post-operative healing and/or osseointegration
* Need for systemic corticosteroids or any other medication that would compromise post-operative healing and/or osseointegration
* History of radiation in the head and neck region
* History of chemotherapy within 5 years prior to surgery
* Unable or unwilling to return for follow-up visits for a period of 3 years and 6 months
* Unrealistic esthetic demands
* Unlikely to be able to comply with study procedures according to Investigators judgement
* Involvement in the planning and conduct of the study (applies to both Astra Tech staff or staff at the investigational site)
* Previous enrolment in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2005-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06-14 (Actual)

PRIMARY OUTCOMES:
Clinical measure of the thickness of the facial bone wall. | At implant placement and after 16 weeks of healing.

CONTACTS AND LOCATIONS:
Locations (3):
- Studio Odontoiatrico, Padua, Italy
- Department of Periodontics, Faculty of Odontology, Universidad Complutense de Madrid, Madrid, Spain
- Department of Periodontology, School of Dental Medicine, University of Berne, Bern, Switzerland

REFERENCES:
- [Result] Huynh-Ba G, Pjetursson BE, Sanz M, Cecchinato D, Ferrus J, Lindhe J, Lang NP. Analysis of the socket bone wall dimensions in the upper maxilla in relation to immediate implant placement. Clin Oral Implants Res. 2010 Jan;21(1):37-42. doi: 10.1111/j.1600-0501.2009.01870.x. PMID 20070745
- [Result] Tomasi C, Sanz M, Cecchinato D, Pjetursson B, Ferrus J, Lang NP, Lindhe J. Bone dimensional variations at implants placed in fresh extraction sockets: a multilevel multivariate analysis. Clin Oral Implants Res. 2010 Jan;21(1):30-6. doi: 10.1111/j.1600-0501.2009.01848.x. PMID 20070744
- [Result] Sanz M, Cecchinato D, Ferrus J, Pjetursson EB, Lang NP, Lindhe J. A prospective, randomized-controlled clinical trial to evaluate bone preservation using implants with different geometry placed into extraction sockets in the maxilla. Clin Oral Implants Res. 2010 Jan;21(1):13-21. doi: 10.1111/j.1600-0501.2009.01824.x. Epub 2009 Nov 18. PMID 19922492
- [Result] Ferrus J, Cecchinato D, Pjetursson EB, Lang NP, Sanz M, Lindhe J. Factors influencing ridge alterations following immediate implant placement into extraction sockets. Clin Oral Implants Res. 2010 Jan;21(1):22-9. doi: 10.1111/j.1600-0501.2009.01825.x. Epub 2009 Nov 13. PMID 19912273
- [Result] Sanz M, Cecchinato D, Ferrus J, Salvi GE, Ramseier C, Lang NP, Lindhe J. Implants placed in fresh extraction sockets in the maxilla: clinical and radiographic outcomes from a 3-year follow-up examination. Clin Oral Implants Res. 2014 Mar;25(3):321-327. doi: 10.1111/clr.12140. Epub 2013 Feb 25. PMID 23431960
- [Result] Cecchinato D, Lops D, Salvi GE, Sanz M. A prospective, randomized, controlled study using OsseoSpeed implants placed in maxillary fresh extraction socket: soft tissues response. Clin Oral Implants Res. 2015;26(1):20-7. doi: 10.1111/clr.12295. Epub 2013 Dec 2. PMID 24298982